CLINICAL TRIAL: NCT01488578
Title: Postmarketing Observational Study of Tolterodine Treatment on Overactive Bladder in Real Life Setting
Brief Title: Tolterodine Drug Use Investigation.(Post Marketing Commitment Plan)
Acronym: POTTOR
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6121186
Record Dates: First submitted 2011-04-27; First posted 2011-12-08 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Japanese; Tolterodine; Detrusitol; Detrol; Postmarketing commitment plan.
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tolterodine tartrate.: Subjects taking Tolterodine tartrate.
  Interventions: Drug: Tolterodine tartrate

INTERVENTIONS:
Drug: Tolterodine tartrate — Detrusitol Capsule 2mg and 4mg, depending on the Investigator prescription.Frequency and duration are according to Package Insert as follows.
  Other Names: Detrusitol Capsule,Tolterodine tartrate.

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the Package Insert (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the subjects whom an investigator prescribes the first Detrusitol Capsule should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects intend to treat their overactive bladder who are prescribed Detrusitol Capsule by their physicians.

Exclusion Criteria:

* Subjects who have been prescribed Detrusitol Capsule before.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects whom an investigator involving A6121186 prescribes the Tolterodine tartrate (Detrusitol Capsule).
Sampling Method: Probability Sample
Enrollment: 11157 (Actual)
Dates: Start 2006-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121186&StudyName=Tolterodine%20drug%20use%20Investigation.%28post%20marketing%20committement%20plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolterodine Tartrate: Participants taking Tolterodine tartrate.
Period: Overall Study
Arm/Group | Tolterodine Tartrate
Started | 11157
Completed | 9321
Not Completed | 1836
Not completed — Protocol Violation | 1836

BASELINE CHARACTERISTICS:
Groups:
- Tolterodine Tartrate: Participants taking Tolterodine tartrate according to Japanese Package Insert.
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 9321
Age, Customized [Number; unit: participants]
  <65 years | 2848
  >=65 years | 6473
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5263
  Male | 4058
Target disease severity [Number; unit: participants] — The severity of Overactive Bladder which was diagnosed by investigator.
  participants
    Mild | 3530
    Moderate | 5185
    Severe | 606
Complications [Number; unit: participants]
  Present | 5837
  Absent | 3484
Concomitant drug [Number; unit: participants]
  Present | 5057
  Absent | 4246
Starting dose [Number; unit: participants]
  2 mg | 1813
  4 mg | 7506
  8 mg | 2

OUTCOME MEASURES:

1. Primary Outcome: Confirmation of the Incidence of All Treatment Related Adverse Events (TRAEs).
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: 12 weeks
Population: Safety analysis population included all enrolled subjects who had received at least 1 confirmed, administration of Detrusitol.
Measure: Number; unit: participants
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 9321
participants | 984

2. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Concomitant Drugs
Description: Number of participants with responders of tolterodine to determine whether with or without concomitant drugs is significant risk factor.
Time Frame: 12 week
Population: The efficacy analysis population consists of the evaluable cases in accordance with the analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Groups:
- With Concomitant Drugs: Participants with concomitant drugs who took tolterodine according to Japanese Package Insert.
- Without Concomitant Drugs: Participants without concomitant drugs who took tolterodine according to Japanese Package Insert.
Arm/Group | With Concomitant Drugs | Without Concomitant Drugs
Number analyzed (Participants) | 4214 | 3566
participants | 3483 | 3053
Statistical Analysis 1: Comparison: With Concomitant Drugs vs Without Concomitant Drugs; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Primary Outcome: Number of Participants Which Was Evaluated as "Degree of Satisfaction".
Description: Participant satisfaction was evaluated by investigators based on questioning the participants at the end of observation period using choices: Satisfied, Dissatisfied, Neither of the above.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 7780
participants
  Satisfied | 5609
  Dissatisfied | 1033
  Neither of the above | 963
  Unknown | 175

4. Primary Outcome: Number of Participants With an Investigator's Assessment of Clinical Outcome at End of the Study.
Description: Clinical overall effectiveness was evaluated by investigators based on clinical symptoms, etc, at the end of observation period.
Time Frame: 12 week
Population: The efficacy analysis population included all subjects from the safety analysis population in whom the efficacy of this drug could be evaluated.
  Number of participants evaluable for which was evaluated "effect".
Measure: Number; unit: participants
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 7780
participants
  Effective | 6536
  Not effective | 1244

5. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Non-drug Therapies
Description: Number of participants with responders of tolterodine to determine whether with or without Non-drug therapies is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Non-drug Therapies: Participants with non-drug therapies who took tolterodine according to Japanese Package Insert.
- Without Non-drug Therapies: Participants without non-drug therapies who took tolterodine according to Japanese Package Insert.
Arm/Group | With Non-drug Therapies | Without Non-drug Therapies
Number analyzed (Participants) | 360 | 7420
participants | 317 | 6219
Statistical Analysis 1: Comparison: With Non-drug Therapies vs Without Non-drug Therapies; Test type: Superiority or Other; p = 0.032, Chi-squared

6. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Gender
Description: Number of participants with responders of tolterodine to determine whether male or female is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Male: Male participants who took tolterodine according to Japanese Package Insert.
- Female: Female participants who took tolterodine according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 3394 | 4386
participants | 2745 | 3791
Statistical Analysis 1: Comparison: Male vs Female; Test type: Superiority or Other; p < 0.001, Chi-squared

7. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Complications
Description: Number of participants with responders of tolterodine to determine whether with or without complications is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Complications: Participants with complications who took tolterodine according to Japanese Package Insert.
- Without Complications: Participants without complications who took tolterodine according to Japanese Package Insert.
Arm/Group | With Complications | Without Complications
Number analyzed (Participants) | 4806 | 2974
participants | 3960 | 2576
Statistical Analysis 1: Comparison: With Complications vs Without Complications; Test type: Superiority or Other; p < 0.001, Chi-squared

8. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Age
Description: Number of participants with responders of tolterodine to determine whether <65 years or >=65 years is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- <65 Years: Participants with < 65 years who took tolterodine according to Japanese Package Insert.
- >=65 Years: Participants with >= 65 years who took tolterodine according to Japanese Package Insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 2379 | 5401
participants | 2060 | 4476
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Tolterodine - Comorbidity of Prostatic Hypertrophy
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of tolterodine to determine whether with or without comorbidity of benign prostatic hypertrophy (BPH) is significant risk factor.
Time Frame: 12 week
Population: The safety analysis population consists of the cases that satisfy the participants conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Groups:
- With BPH: Participants with complication of benign prostatic hypertrophy who took tolterodine according to Japanese Package Insert.
- Without BPH: Participants without complication of benign prostatic hypertrophy who took tolterodine according to Japanese Package Insert.
Arm/Group | With BPH | Without BPH
Number analyzed (Participants) | 2203 | 1855
participants | 319 | 130
Statistical Analysis 1: Comparison: With BPH vs Without BPH; Test type: Superiority or Other; p < 0.001, The Hosmer-Lemeshow Goodness-of-Fit TEST

10. Secondary Outcome: Number of Unlisted Treatment Related Adverse Events (TRAEs)Reported in at Least 5 Participants
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: 12 week
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 9321
events
  Abdominal discomfort | 18
  Pollakiuria | 11
  Cystitis | 10
  Abdominal distension | 10
  Pruritus | 6
  Stomatitis | 5
  Malaise | 5

11. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Severity of Overactive Bladder
Description: Number of participants with responders of tolterodine to determine whether mild, moderate or severe is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Mild: Participants with mild OAB who took tolterodine according to Japanese Package Insert.
- Moderate: Participants with moderate OAB who took tolterodine according to Japanese Package Insert.
- Severe: Participants with severe OAB who took tolterodine according to Japanese Package Insert.
Arm/Group | Mild | Moderate | Severe
Number analyzed (Participants) | 2896 | 4378 | 506
participants | 2426 | 3709 | 401
Statistical Analysis 1: Comparison: Mild vs Moderate vs Severe; Test type: Superiority or Other; p = 0.006, Chi-squared

12. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Urinary Urgency
Description: Number of participants with responders of tolterodine to determine whether with or without Urinary urgency is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Urinary Urgency: Participants with urinary urgency who took tolterodine according to Japanese Package Insert.
- Without Urinary Urgency: Participants without urinary urgency who took tolterodine according to Japanese Package Insert.
Arm/Group | With Urinary Urgency | Without Urinary Urgency
Number analyzed (Participants) | 6521 | 1043
participants | 5529 | 829
Statistical Analysis 1: Comparison: With Urinary Urgency vs Without Urinary Urgency; Test type: Superiority or Other; p < 0.001, Chi-squared

13. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Number of Urinations Per Day (During Sleep)
Description: Number of participants with responders of tolterodine to determine the Number of urinations per day (during sleep) is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- No Urination: Participants with no urination who took tolterodine according to Japanese Package Insert.
- 1 Urination: Participants with 1 time urination per day (during sleep)who took tolterodine according to Japanese Package Insert.
- 2 Urinations: Participants with 2 times urination per day (during sleep)who took tolterodine according to Japanese Package Insert.
- >= 3 Urinations: Participants with >= 3 times urination per day (during sleep)who took tolterodine according to Japanese Package Insert.
Arm/Group | No Urination | 1 Urination | 2 Urinations | >= 3 Urinations
Number analyzed (Participants) | 442 | 1021 | 1600 | 4223
participants | 370 | 882 | 1380 | 3523
Statistical Analysis 1: Comparison: No Urination vs 1 Urination vs 2 Urinations vs >= 3 Urinations; Test type: Superiority or Other; p = 0.015, Chi-squared

14. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Number of Urinary Incontinence Episodes Per Day
Description: Number of participants with responders of tolterodine to determine the Number of urinary incontinence episodes per day is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- 1 to 2 Episodes: Participants with 1 or 2 urinary incontinence episodes per day who took tolterodine according to Japanese Package Insert.
- 3 to 4 Episodes: Participants with 3 or 4 urinary incontinence episodes per day who took tolterodine according to Japanese Package Insert.
- >= 5 Episodes: Participants with >= 5 urinary incontinence episodes per day who took tolterodine according to Japanese Package Insert.
Arm/Group | 1 to 2 Episodes | 3 to 4 Episodes | >= 5 Episodes
Number analyzed (Participants) | 1913 | 836 | 322
participants | 1670 | 710 | 254
Statistical Analysis 1: Comparison: 1 to 2 Episodes vs 3 to 4 Episodes vs >= 5 Episodes; Test type: Superiority or Other; p < 0.001, Chi-squared

15. Secondary Outcome: Risk Factors for the Proportion of Responders of Tolterodine-Previous Treatment
Description: Number of participants with response to tolterodine to determine whether with or without previous treatment is significant risk factor.
Time Frame: 12 week
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Previous Treatment: Participants with previous treatment of OAB who took tolterodine according to Japanese Package Insert.
- Without Previous Treatment: Participants without previous treatment of OAB who took tolterodine according to Japanese Package Insert.
Arm/Group | With Previous Treatment | Without Previous Treatment
Number analyzed (Participants) | 943 | 6736
participants | 698 | 5753
Statistical Analysis 1: Comparison: With Previous Treatment vs Without Previous Treatment; Test type: Superiority or Other; p < 0.001, Chi-squared

16. Primary Outcome: Confirmation of Frequent Treatment Related Adverse Events (TRAEs) at the End of Observation Period.
Description: The Treatment Related Adverse Events (TRAEs) at the end of observation period with an incidence of 1% or higher.
Time Frame: 12 week
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Tolterodine Tartrate
Number analyzed (Participants) | 9321
events
  Thirst | 344
  Constipation | 194
  Dysuria | 166

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tolterodine Tartrate
Serious Adverse Events (participants affected / at risk) | 12/9321
Other Adverse Events (participants affected / at risk) | 703/9321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine Tartrate (N=9321)
Urinary retention (Renal and urinary disorders) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine Tartrate (N=9321)
Thirst (General disorders) | 344 (344)
Constipation (Gastrointestinal disorders) | 194 (194)
Dysuria (Renal and urinary disorders) | 165 (165)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.